CLINICAL TRIAL: NCT02379910
Title: AM1030: A Phase I/II, Double-Blind, Placebo-Controlled, Single and Multiple Ascending (Topical) Dose, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Study in Patients (Male and Female) With Atopic Dermatitis
Brief Title: A Study to Assess the Safety, Tolerability, PK and PD of AM1030-CREAM in Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AnaMar AB (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1030-260-01; 2014-003684-38 (EudraCT Number)
Record Dates: First submitted 2015-02-19; First posted 2015-03-05 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- SAD 1 (Experimental): AM1030-CREAM
  Interventions: Drug: AM1030-CREAM or placebo
- SAD 2 (Experimental): AM1030-CREAM
  Interventions: Drug: AM1030-CREAM or placebo
- SAD 3 (Experimental): AM1030-CREAM
  Interventions: Drug: AM1030-CREAM or placebo
- MAD 1 (Experimental): AM1030-CREAM
  Interventions: Drug: AM1030-CREAM or placebo
- MAD 2 (Experimental): AM1030-CREAM
  Interventions: Drug: AM1030-CREAM or placebo

INTERVENTIONS:
Drug: AM1030-CREAM or placebo

SUMMARY:
This is a study of safety, tolerability, pharmacokinetics and pharmacodynamics of AM1030-CREAM in patients with Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females of any ethnic origin between 18 and 65 years of age
* Body mass index between 18.0 and 35.0 kg/m2
* Subjects with AD as defined by the Hanifen and Rajka criteria and with mild to severe disease activity (IGA 2-4)
* AD lesions amenable to cutaneous treatment located on the trunk and/or limbs

Exclusion Criteria:

* Subjects with scars, moles, tattoos, sunburn or other blemishes in test areas
* Systemic treatment with immunosuppressants, immunomodulators or corticosteroids within 2 weeks prior to dosing
* Topical treatment with corticosteroids, antibiotics and/or immunomodulators within 4 days prior to dosing
* Treatment with systemic antihistamines within 24 hours of the first dose administration
* Treatment with SSRIs within 2 weeks of the first dose administration
* Subjects who have received phototherapy within 4 weeks prior to dosing

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Day 1-15
  Number of adverse events as a measure of Safety
Local Tolerability: Change in Erythema (Likert scale 0-4) | Day 1-15
  Change in Erythema (Likert scale 0-4) as a measure of Local Tolerability
Local Tolerability: Change in Oedema (Likert scale 0-3) | Day 1-15
  Change in Oedema (Likert scale 0-3) as a measure of Local Tolerability
Local Tolerability: Change in Burning (Likert scale 0-3) | Day 1-15
  Change in Burning (Likert scale 0-3) as a measure of Local Tolerability
Local Tolerability: Change in Prutitus (VAS) | Day 1-15
  Change in Prutitus (VAS) as a measure of Local Tolerability
Vital Signs | Day 1-15
  Change in blood pressure as a measure of Safety
Vital Signs | Day 1-15
  Change in pulse rate as a measure of Safety
Vital Signs | Day 1-15
  Change in body temperature as a measure of Safety
ECG | Day 1-15
  Change in ECG as a measure of Safety
Physical Examination | Day 1-15
  Any abnormal observations from Physical Examination as a measure of Safety

SECONDARY OUTCOMES:
Pharmacokinetics: Cmax, AUC, tmax, t1/2, Vss/F, CL/F | Profil Day 1-15
  Pharmacokinetics as measured by Cmax, AUC, tmax, t1/2, Vss/F, CL/F
Pruritus on a Visual Analog Scale | Day 1-15
  Pruritus (Visual Analog Scale 10 cm) as a measure of Efficacy
Erythema on a Likert scale | Day 1-15
  Erythema (Likert Scale 0-4) as a measure of Efficacy
Modified Eczema Area and Severity Index (mEASI) | Day 1-15
  mEASI (Composite score 0-64.8) as a measure of Efficay

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, Principal Investigator — Covance CRU
Locations (2):
- United Kingdom (2):
  - Covance CRU, Leeds
  - CRLCRU Royal Liverpool University Hospital, Liverpool